CLINICAL TRIAL: NCT06024902
Title: Clinical Characteristics of Severe Childhood Asthma
Status: Completed | Type: Observational
Sponsor: Children's Hospital of Fudan University (Other)
Responsible Party: Sponsor
Other Study IDs: 2023-002
Record Dates: First submitted 2023-08-30; First posted 2023-09-06 (Actual); Last update posted 2023-12-22 (Actual); Status verified 2023-12

CONDITIONS: Severe Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- childhood asthma: Subjects with confirmed diagnosis of asthma without other lung disease followed for collection of demographic and clinical data.

SUMMARY:
Asthma remains a serious health problem with increasing prevalence and incidence. There is limited information about severe asthma among Chinese pediatric patients. In this context, we decided to explore the clinical characteristics and risk factors of severe asthma in children. This is a descriptive, observational, retrospective cohort study in children with asthma.

The purpose of this retrospective study is: to determine the clinical characteristics of severe asthma of children; to identify the factors associated with severe childhood asthma.

DETAILED DESCRIPTION:
Asthma remains a serious health problem with increasing prevalence and incidence. There is limited information about severe asthma among Chinese pediatric patients. In this context, we decided to explore the clinical characteristics and risk factors of severe asthma in children. This is a descriptive, observational, retrospective cohort study in children with asthma.

The purpose of this retrospective study is: to determine the clinical characteristics of severe asthma of children; to identify the factors associated with severe childhood asthma.

Participants were consecutively recruited from asthma clinics between January 2021 and December 2021 at Children's Hospital of Fudan University. Patients fulfilling the following criteria were eligible for inclusion: (1) aged 6-17 years old; (2) diagnosed with asthma according to the Global Initiative for Asthma (GINA) 2020 guideline; (3) children and their caregivers are informed and voluntarily join the database and had follow up for at least 1 year. Patients who had cystic fibrosis, mechanical airway obstruction, or any other pulmonary disease or whose parents or legal guardians were not able to fill in the questionnaires were not enrolled.

At baseline, the asthma specialist questioned each of the patient in the presence of their caregivers to ensure that they supplied accurate disease information and were included according to the criteria. The patients and their caregivers are asked to complete the online questionnaires including the demographic; baseline asthma control, triggers, exacerbation, medication and adherence; environmental exposure, and diagnosis and control of comorbidities, etc. If a patient had poorly controlled comorbidities, multidisciplinary consultation would be recommended. Clinical assessments were arranged at baseline, 3, 6, 9, and 12 months.

ELIGIBILITY:
Inclusion Criteria:

* (1) aged 6-17 years old;
* (2) diagnosed with asthma according to the Global Initiative for Asthma (GINA) 2020 guideline;
* (3) children and their caregivers are informed and voluntarily join the database and had follow up for at least 1 year.

Exclusion Criteria:

* (1) Patients with cystic fibrosis;
* (2) had mechanical airway obstruction, or any other pulmonary disease;
* (3) whose parents or legal guardians were not able to fill in the questionnaires.

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: The tertiary specialized children's hospital
Sampling Method: Non-Probability Sample
Enrollment: 650 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Severity of asthma | 12 months
  The severity of asthma was comprehensively estimated by a pediatric pulmonologist following the criteria of the Global Initiative for Asthma (GINA) 2021(collecting clinical characteristics, questionnaires and Pulmonary function tests)when patients completed 12-months management.

CONTACTS AND LOCATIONS:
Locations (1):
- Children's Hospital of Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No